CLINICAL TRIAL: NCT02684942
Title: Comparison of Meperidine and Fentanyl on Pain Scale and Quality of Life in Cervical Cancer Patients Receiving Brachytherapy: A Double-blind, Randomized Controlled Trial
Brief Title: Comparison of Meperidine and Fentanyl on Pain Scale and QOL in Brachytherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulabhorn Cancer Center (Other)
Responsible Party: Principal Investigator, Saengrawee Thanthong, Mrs, OCN, Chulabhorn Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20/2553
Record Dates: First submitted 2016-01-29; First posted 2016-02-18 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Pain; Quality of Life
Keywords: Meperidine; Fentanyl; Pain management; brachytherapy
MeSH Terms: conditions — Pain; Agnosia | interventions — Meperidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Meperidine,Fentanyl,Meperidine,Fentanyl (Active Comparator): Injection meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at first and third fraction of brachytherapy. And injection fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at second and fourth fraction of brachytherapy.
  Interventions: Drug: Meperidine; Drug: Fentanyl
- Fentanyl,Meperidine,Fentanyl,Meperidine (Active Comparator): Injection meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at second and fourth fraction of brachytherapy. And injection fentanyl 1 umg/kg to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at first and third fraction of brachytherapy.
  Interventions: Drug: Meperidine; Drug: Fentanyl
- Meperidine,Meperidine,Fentanyl,Fentanyl (Active Comparator): Injection meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at first and second fraction of brachytherapy. And injection fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at third and fourth fraction of brachytherapy.
  Interventions: Drug: Meperidine; Drug: Fentanyl
- Fentanyl,Fentanyl,Meperidine,Meperidine (Active Comparator): Injection meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at third and fourth fraction of brachytherapy. And injection fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at first and second fraction.
  Interventions: Drug: Meperidine; Drug: Fentanyl
- Meperidine,Fentanyl,Fentanyl,Meperidine (Active Comparator): Injection meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at first and fourth fraction of brachytherapy. And injection fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score more than 4 at second and third fraction of brachytherapy.
  Interventions: Drug: Meperidine; Drug: Fentanyl
- Fentanyl,Meperidine,Meperidine,Fentanyl (Active Comparator): Injection meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at second and third fractionof brachytherapy. And injection fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4 at first and fourth fraction of brachytherapy.
  Interventions: Drug: Meperidine; Drug: Fentanyl

INTERVENTIONS:
Drug: Meperidine — Injection meperidine 1 mg/kg with diazepam 0.1 mg/kg.to intravenous 5 minutes before inserting the applicator and then when the patients had pain score greater or equal to 4. All patients received supplement oxygen cannula 3 LPM continuously monitored for saturation, pulse and monitored every 5 minutes for blood pressure.
  Other Names: Pethidine
Drug: Fentanyl — Injection meperidine 1 mg/kg to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4. All patients received supplement oxygen cannula 3 LPM continuously monitored for saturation, pulse and monitored every 5 minutes for blood pressure.
  Other Names: Fentanil

SUMMARY:
Purpose: To compare the pain level and quality of life of the two sedation regimens consisting of diazepam in combination with meperidine or fentanyl.

Materials and methods: A total of 40 patients (160 sessions of brachytherapy), unselected brachytherapy out patients at Chulabhorn Hospital, Thailand were enrolled with informed consent and randomized to receive meperidine or fentanyl. Data of perceived pain (according to standard 10-cm visual analog scales [VAS]), and perceived Quality of life (EQ-5D) were collected. Patients and all brachytherapy staffs directly involved with the procedure were blinded about the drug used.

DETAILED DESCRIPTION:
Methods Patients Unselected, forty female adults, aged 20 years old or older, diagnosed with cervical cancer and treated with brachytherapy as outpatients at Chulabhorn Hospital, Thailand between June 2011 and September 2012 were enrolled in the study with their informed consents. The study was approved by The Chulabhorn Research Institutional Review Board and Chulabhorn Ethics committee. All the patients were treated with four sessions of ICRT(Intracavitary Radiation Therapy). Inclusion criteria were: Age 20 - 80 years, can understand and provide information, no trouble hearing and good conscious, agree to participated and had performance levels at ECOG 0-2. The patients were randomized to receive either meperidine (1 mg/kg) or fentanyl (1 ug/kg) with diazepam 10 mg both. Nursing staffs who prepared the drugs picked the drugs from lotteries organized into 6 lots on it.

Procedures Perceived pain score according to standard 10-cm visual analog scales (VAS) was assessed prior to treatment and every 15 minutes from the start to the end of the ICRT procedure. Perceived Quality of life (EQ-5D) was assessed before the treatment and immediately after the completion of each brachytherapy treatment session. Information regarding which drug was used was concealed to all the patients and brachytherapy staffs directly involved with the procedures. The procedures involved a radiation oncologist, two nurses, a practical nurse, a radiotherapist, and a medical physicist.

Firstly, before the procedure the patients must NPO(Nothing per oral) for 6 hours and was inserted with intravenous catheter for IV sedation drug depending on the randomized drug that they received.

Secondly, the patients laid down on brachytherapy stretcher and were treated according to the standard ICRT protocol. Each randomized patient had 4 fractions of ICRT, so a single patient will receive Fentanyl and Diazepam 2 fractions and Meperidine and Diazepam 2 fractions. The drugs used were diluted with normal saline to 10 ml. and labeled as "Protocol drug". The actual content within the syringes was known only to a nurse that did not directly involve in the study. Syringes prepared for the meperidine group contained 50 mg of meperidine, while syringes prepared for the fentanyl group contained 100 mg of fentanyl. Both drugs were drawn into 10-cc syringes and appeared colorless.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years old or older,
* Diagnosed with cervical cancer
* On course of external Radiation therapy
* Treated with brachytherapy 4 times.

Exclusion Criteria:

* Pregnant
* Previously underwent intracavitary brachytherapy
* Illiterate

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saengrawee Thanthong, RN., Principal Investigator — 54 moo 4 Kampangpet 6 Taladbangken Laksi Bangkok, THAILAND 10210

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Davidson SE, Symonds RP, Lamont D, Watson ER. Does adenocarcinoma of uterine cervix have a worse prognosis than squamous carcinoma when treated by radiotherapy? Gynecol Oncol. 1989 Apr;33(1):23-6. doi: 10.1016/0090-8258(89)90596-9. PMID 2495240
- [Background] Arunachalam D, Thirumoorthy A, Devi S, Thennarasu. Quality of Life in Cancer Patients with Disfigurement due to Cancer and its Treatments. Indian J Palliat Care. 2011 Sep;17(3):184-90. doi: 10.4103/0973-1075.92334. PMID 22346042
- [Background] Dzeletovic I, Harrison ME, Crowell MD, Ramirez FC, Yows CR, Harris LA, Pasha SF, Gurudu SR, Leighton JA, Heigh RI. Impact of fentanyl in lieu of meperidine on endoscopy unit efficiency: a prospective comparative study in patients undergoing EGD. Gastrointest Endosc. 2013 Jun;77(6):883-7. doi: 10.1016/j.gie.2013.01.013. Epub 2013 Mar 6. PMID 23472999
- [Background] Patel NC, Heckman MG, Palmer WC, Cangemi D, DeVault KR. A comparison of patient satisfaction with sedation between fentanyl/midazolam and meperidine/midazolam in patients undergoing endoscopy. Am J Gastroenterol. 2014 May;109(5):772-4. doi: 10.1038/ajg.2014.31. No abstract available. PMID 24797008
- [Background] Kwekkeboom KL, Dendaas NR, Straub M, Bradley KA. Patterns of pain and distress during high-dose-rate intracavity brachytherapy for cervical cancer. J Support Oncol. 2009 May-Jun;7(3):108-14. PMID 19507459
- [Background] Movafegh A, Ghafouri A, Nasr-Esfahani M, Gholamrezanezhad A, Madhkhan S. Post-thoracotomy analgesia--comparison epidural fentanyl to intravenous pethidine. Middle East J Anaesthesiol. 2007 Feb;19(1):111-22. PMID 17511187
- [Background] Robertson DJ, Jacobs DP, Mackenzie TA, Oringer JA, Rothstein RI. Clinical trial: a randomized, study comparing meperidine (pethidine) and fentanyl in adult gastrointestinal endoscopy. Aliment Pharmacol Ther. 2009 Apr 15;29(8):817-23. doi: 10.1111/j.1365-2036.2009.03943.x. Epub 2009 Jan 20. PMID 19154568
- [Background] Smith MD, Todd JG, Symonds RP. Analgesia for pelvic brachytherapy. Br J Anaesth. 2002 Feb;88(2):270-6. doi: 10.1093/bja/88.2.270. PMID 11878659
- [Background] Soysal S, Karcioglu O, Demircan A, Topacoglu H, Serinken M, Ozucelik N, Tirpan K, Gunerli A. Comparison of meperidine plus midazolam and fentanyl plus midazolam in procedural sedation: a double-blind, randomized controlled trial. Adv Ther. 2004 Sep-Oct;21(5):312-21. doi: 10.1007/BF02850035. PMID 15727400
- [Result] Agostoni M, Fanti L, Arcidiacono PG, Gemma M, Strini G, Torri G, Testoni PA. Midazolam and pethidine versus propofol and fentanyl patient controlled sedation/analgesia for upper gastrointestinal tract ultrasound endoscopy: a prospective randomized controlled trial. Dig Liver Dis. 2007 Nov;39(11):1024-9. doi: 10.1016/j.dld.2007.08.004. Epub 2007 Oct 29. PMID 17913605
- [Derived] Thanthong S, Rojthamarat S, Worasawate W, Vichitvejpaisal P, Nantajit D, Ieumwananontachai N. Comparison of efficacy of meperidine and fentanyl in terms of pain management and quality of life in patients with cervical cancer receiving intracavitary brachytherapy: a double-blind, randomized controlled trial. Support Care Cancer. 2017 Aug;25(8):2531-2537. doi: 10.1007/s00520-017-3662-3. Epub 2017 Mar 18. PMID 28315010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study design is cross-over in female outpatients with cervical cancer (age, 20-80 years) stage IB-IVB treated with four fractions of brachytherapy from June 2013 to September 2014 were enrolled in the study.
Pre-assignment Details: Forty patients with cervical cancer were enrolled in the study. The exclusion criteria were prior pelvic brachytherapy and a history of allergy to meperidine, fentanyl, or benzodiazepine and none were subsequently excluded.
Groups:
- Meperidine,Fentanyl,Meperidine,Fentanyl: First and Third Intervention inject meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
  Second and Fourth Intervention inject fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
- Fentanyl,Meperidine,Fentanyl,Meperidine: First and Third Intervention inject inject fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
  Second and Fourth Intervention inject meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
- Meperidine,Meperidine,Fentanyl,Fentanyl: First and Second Intervention inject meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
  Third and Fourth Intervention inject fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
- Fentanyl,Fentanyl,Meperidine,Meperidine: First and Second Intervention inject fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
  Third and Fourth Intervention inject meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
- Meperidine,Fentanyl,Fentanyl,Meperidine: First and Fourth Intervention inject meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
  Second and Third Intervention inject fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
- Fentanyl,Meperidine,Meperidine,Fentanyl: First and Fourth Intervention inject fentanyl 1 ug./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
  Second and Third Intervention inject meperidine 1 mg./kg. to intravenous 5 minute before insertion the applicator and then when the patients had pain score greater than or equal to 4.
Period: Overall Study
Arm/Group | Meperidine,Fentanyl,Meperidine,Fentanyl | Fentanyl,Meperidine,Fentanyl,Meperidine | Meperidine,Meperidine,Fentanyl,Fentanyl | Fentanyl,Fentanyl,Meperidine,Meperidine | Meperidine,Fentanyl,Fentanyl,Meperidine | Fentanyl,Meperidine,Meperidine,Fentanyl
Started | 7 | 7 | 7 | 7 | 6 | 6
Completed | 7 | 7 | 7 | 7 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who enrolled to this study.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Study in patients with cervical cancer.
  Participants
    Female | 40
    Male | 0
Radiation modality [Number; unit: participants] — Generally, the brachytherapy technique divided into two methods; 1.2D method is based on 2D imaging x-ray 2.3D method is based on 3D imaging which have been incorporated into treatment planning methods, allowing full 3D dose distributions to be computed.
  participants
    2D, two-dimensional | 30
    3D conformal | 10
FIGO stage [Number; unit: participants] — Cervical cancer staging at diagnosis was based on the International Federation of Gynecology and Obstetrics (FIGO).
  Stage I is the least severe, where the tumor is confined to the cervix. Stage II Tumor invades beyond uterus but not to pelvic wall or lower third of vagina.
  Stage III Extends to pelvic wall and/or lower 1/3 vagina and/or causes hydronephrosis or nonfunctional kidney.
  Stage IV Is the most severe, Tumor invades mucosa of bladder or rectum and/or extends beyond true pelvis.
  participants
    IB | 5
    IIA1 | 2
    IIA2 | 1
    IIB | 16
    IIIB | 15
    IVB | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Perceived pain score according to standard 10-cm visual analog scales (VAS) was assessed before injection of medicine for every 15 minutes up to 120 minutes.The minimum and maximum scores were 0, 10. Score 0 means no pain, 1-3 mild pain, 4-6 moderate pain, 7-9 severe pain and 10 worst pain.
Time Frame: From date of the first fraction until date of the last fraction of brachytherapy, once a week for four weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: fraction
Groups:
- Meperidine: Separate analysis in meperidine group.
- Fentanyl: Separate analysis in fentanyl group.
Arm/Group | Meperidine | Fentanyl
Number analyzed (Participants) | 40 | 40
Number analyzed (fraction) | 80 | 80
units on a scale
  baseline | 0.04 (0.25) | 0.14 (0.55)
  0 minute | 0.49 (1.18) | 0.40 (1.16)
  15 minute | 0.59 (1.38) | 0.65 (1.21)
  30 minute | 1.05 (1.76) | 1.24 (2.21)
  45 minute | 1.33 (2.09) | 1.70 (2.48)
  60 minute | 0.61 (1.48) | 0.81 (1.83)
  75 minute | 0.49 (0.99) | 0.53 (1.12)
  90 minute | 0.24 (0.80) | 0.13 (0.58)
  105 minute | 0.24 (0.80) | 0.13 (0.58)
  120 minute | 0.24 (0.80) | 0.13 (0.58)

2. Secondary Outcome: Quality of Life
Description: Perceived Quality of life (EQ-5D) was assessed before the first brachytherpy and immediately after completion of each of the 4 brachytherapy fractions. The EQ-5D have 5 dimensions: mobility, self-care, usual activities, topics each content 3 responses: no problems, some problems, extreme problems.
Time Frame: From date of the first fraction of brachytherapy until date of the last fraction of brachytherapy,once a week for 4 weeks
Population: Pain score in each fraction.
Measure: Number; unit: participants
Units Other Than Participants: fraction
Groups:
- Meperidine: Separate analyze in fraction that patient receive meperidine.
- Fentanyl: Separate analyze in fraction that patient received fentanyl.
Arm/Group | Meperidine | Fentanyl
Number analyzed (Participants) | 40 | 40
Number analyzed (fraction) | 80 | 80
participants
  No problems in mobility | 62 | 58
  Some problems in mobility | 16 | 18
  Severe problems in mobility | 1 | 1
  No problem in self-care | 68 | 69
  Some problem in self-care | 11 | 6
  Severe problem in self-care | 0 | 2
  No problem in usual activities | 55 | 53
  Some problem in usual activities | 22 | 21
  Severe problem in usual activities | 2 | 3
  No problem in pain/discomfort | 27 | 23
  Some problem in pain/discomfort | 49 | 53
  Severe problem in pain/discomfort | 3 | 1
  No problem in anxiety/depression | 46 | 42
  Some problem in anxiety/depression | 32 | 33
  Severe problem in anxiety/depression | 1 | 2

3. Other Pre Specified Outcome: Ovoids Size
Description: Size of ovoids that a pair part of brachytherapy applicator insert in vagina trough cervix.
Time Frame: after complete applicator insertion.
Population: Each patient was treated with 4 fractions of brachytherapy.
Measure: Median (Full Range); unit: Centimeter
Units Other Than Participants: fraction
Groups:
- Meperidine: Analyze in meperidine group.
- Fentanyl: Analyze in fentanyl group.
Arm/Group | Meperidine | Fentanyl
Number analyzed (Participants) | 40 | 40
Number analyzed (fraction) | 80 | 80
Centimeter | 2 [1.5 to 3] | 2 [1.5 to 3]

4. Other Pre Specified Outcome: Tumor Size
Description: Size of tumor at cervix measured by the doctor before insert applicator.
Time Frame: Before insert applicator in each fraction of brachytherapy.
Population: Participants received 4 fraction of brachytherapy. Thus all 160 fractions separated to two group of drug and analysis data in each group.
Measure: Mean (Standard Deviation); unit: CM.
Units Other Than Participants: fraction
Arm/Group | Meperidine | Fentanyl
Number analyzed (Participants) | 40 | 40
Number analyzed (fraction) | 80 | 80
CM. | 2.23 (1.29) | 2.21 (1.25)

5. Other Pre Specified Outcome: Meperidine Dose
Description: Sum of meperidine dose when finish each fraction of brachytherapy
Time Frame: after complete treatment.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg.
Units Other Than Participants: fraction
Arm/Group | Meperidine
Number analyzed (Participants) | 40
Number analyzed (fraction) | 80
mg. | 50.13 (0.26)

6. Other Pre Specified Outcome: Fentanyl Dose
Description: Sum of fentanyl dose when finish each fraction of brachytherapy
Time Frame: after complete treatment.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug.
Units Other Than Participants: fraction
Arm/Group | Fentanyl
Number analyzed (Participants) | 40
Number analyzed (fraction) | 80
ug. | 100.18 (0.32)

ADVERSE EVENTS:
Time Frame: 1-day
Description: Adverse events were monitored throughout each 1-day intervention
Arm/Group | Meperidine | Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No